CLINICAL TRIAL: NCT05397873
Title: Biofeedback Training to Improve Fixation Stability, Visual Function Outcomes, and Quality of Life in Hemianopia Cases
Brief Title: Biofeedback for Hemianopia Vision Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Monica Nido, Associate Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Toronto
Record Dates: First submitted 2021-12-01; First posted 2022-05-31 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Hemianopsia, Homonymous; Brain Injury; Stroke; Brain Tumor; Brain Trauma
Keywords: hemianopsia; stroke; brain tumor; brain trauma; visual fields; visual loss; low vision; fixation stability; biofeedback training; MAIA microperimeter
MeSH Terms: conditions — Hemianopsia; Brain Injuries; Stroke; Brain Neoplasms; Brain Injuries, Traumatic; Vision Disorders; Vision, Low

STUDY DESIGN:
Intervention Model Description: A group of patients have the intervention and another group has control tests.
Who Masked: Outcomes Assessor
Masking Description: The assessor does not know if the patient is in the control group, treatment group or cross over group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The patients will undergo baseline assessment and receive the intervention, being assessed after the intervention.
  Interventions: Device: Biofeedback training
- Group B (No Intervention): The patients will perform the same tests for assessment as in group A, however, no intervention will be done. They may enrol in the study as group B after completing group B participation.

INTERVENTIONS:
Device: Biofeedback training — The training of oculomotor functions is done on the biofeedback module of a microperimeter MAIA.
  Arms: Group A

SUMMARY:
Patients with brain injury secondary to stroke, surgery, or trauma frequently suffer from homonymous hemianopia, defined as vision loss in one hemifield secondary to retro- chiasmal lesion. Classic and effective saccadic compensatory training therapies are current aim to reorganize the control of visual information processing and eye movements or, in other words, to induce or improve oculomotor adaptation to visual field loss. Patients learn to intentionally shift their eyes and, thus, their visual field border, into the area corresponding to their blind visual field. This shift brings the visual information from the blind hemifield into the seeing hemifield for further processing. Patients learn, therefore, to efficiently use their eyes "to keep the 'blind side' in sight". Biofeedback training (BT) is the latest and newest technique for oculomotor control training in cases with low vision when using available modules in the new microperimetry instruments. Studies in the literature highlighted positive benefits from using BT in a variety of central vision loss, nystagmus cases, and others.The purpose of this study is to assess systematically the impact of BT in a series of cases with hemianopia and formulate guidelines for further use of this intervention in vision rehabilitation of hemianopia cases in general.

DETAILED DESCRIPTION:
Background

Patients with brain injury secondary to stroke, surgery, or trauma frequently suffer from homonymous hemianopia, defined as vision loss in one hemifield secondary to retro- chiasmal lesion. About 45% of stroke survivors have homonymous hemianopia. A deficit in vision and spatial perception can cause slowdown of the rehabilitation progress in physiotherapy.

According to Kerkhoff 1patients face three main visual behavioral problems: (1) impaired eye movements (including saccades) leading to defective visual and spatial exploration, (2) hemianopic reading deficit (hemianopic alexia) because of the parafoveal field loss and (3) deviated subjective midline. Hemianopic dyslexia is not simply the product of the visual field defect but is caused by a disorder of control of visual information processing and eye movements in reading.

Most important, the capability to read is fundamental for daily living and an essential prerequisite for education and success in our modern society, so this disorder can have a profound effect on patients' lives. Patients with visual field loss usually fail to adapt to their reading impairment (80% of cases). In these cases, word identification and the abilities to plan and guide reading eye movements are disturbed.

In spite of these facts, visual rehabilitation program on a larger scale is still missing in most rehabilitation centers and clinics. This is decurrent to the generalized belief that lesions of the lateral geniculate nucleus and striate cortex lead to a permanent loss of vision. According to scientific findings, this does not always have to be true.

Classic and effective saccadic compensatory training therapies are current.5 They aim to reorganize the control of visual information processing and eye movements or, in other words, to induce or improve oculomotor adaptation to visual field loss. Such therapies involve the systematic and repetitive practice of specific eye movements for reading or for visual exploration. Patients learn to intentionally shift their eyes and, thus, their visual field border, into the area corresponding to their blind visual field. This shift brings the visual information from the blind hemifield into the seeing hemifield for further processing. Patients learn, therefore, to efficiently use their eyes "to keep the 'blind side' in sight". The training-induced, efficient oculomotor adaptation to visual field loss becomes manifest as a change of reading (or visual exploration) eye-movement patterns and indicates the functional reorganization of the control of visual information processing and eye movements.6

Biofeedback training for active eye movement control was never used in hemianopia cases before. Biofeedback training (BT) is the latest and newest technique for oculomotor control training in cases with low vision when using available modules in the new microperimetry instruments.7-9 Studies in the literature highlighted positive benefits from using BT in a variety of central vision loss, nystagmus cases, and others.10-18 The purpose of this study is to assess systematically the impact of BT in a series of cases with hemianopia and formulate guidelines for further use of this intervention in vision rehabilitation of hemianopia cases in general.

Rationale for the study

The deviation of the subjective midline in hemianopia cases brings visual perception from a line of objects in the surrounds to be at a much higher-level of perception/cognition, thus disturbing reading, gait and balance. Besides that, impaired saccades also cause wrong exploration patterns and deteriorated visual search. It results in the prolonged exploration time of a scene and can lead to significant problems in daily life such as inability to navigate around various obstacles (cars, people and other objects). It also causes a cognitive deficit while extracting information from a visual scene. 1 A combination of factors such as reduced contrast sensitivity, impaired visual search and inaccurate fixation contributes to the matter.

Visual information extraction from the parafoveal visual field provides the basis for planning and guiding of reading eye movements. Therefore, patients with hemianopia have difficulties in shifting their gaze systematically from left to right (in right-sided field loss) or finding the beginning of a new line (in left sided field loss). Such eye movements are optimized by visual feedback. BT promotes luminous and auditory biofeedback, which potentializes its efficacy in vision rehabilitation.

BT in the microperimeter module provides the accurate and efficient oculomotor training necessary to relocate the subjective midline to the seeing field in 1-20 or even more, as needed. BT also improves dramatically fixation stability and saccades. The advantage of this training method over classic training is potentially great. Firstly, the highest retinal sensitivity convenient point can be identified considering the whole visual field. The microperimeter provides real time scrutiny of ocular movements on a screen, and the therapist is able to select precisely the trained retinal locus (FFT) to be used by the patient on top of the microperimeter visual field. Finally, according to the patients' response the FFT can be readjusted. Eight cases trained with BT for hemianopia in our low vision rehabilitation (LVR) service had marked improvements in fixation stability, and microperimeter fields.

Expansion of visual space in the direction of the blind field and compression of visual space in the direction of the seeing field may be a contributory factor to the altered perception of their egocentric directional sense and overall more veridical mapping of their visual space, as well as the resultant shift in their positional centre of gravity. We hypothesize that BT promotes this field relocation.

Conventional visual exploration training studies have confirmed that 10 to 25 training sessions in a 6-week period can be effective for hemianopia patients to adopt these strategies. BT is able to achieve significant results in 5 weekly sessions of 20 minutes each, according to 8 cases treated in our service.

Study hypothesis

The visual and audio parts of the BT program improve in a synergistic way oculomotor control through attention improvement and volitional eye movements towards pre-designated targets. Improved oculomotor control results in better fixation stability of eyes. Better fixation stability in turn results in better navigation for distance and near vision reading. Dual sensory BT is a therapy used in low vision for more than ten years, showing good results for near and distance vision in cases with macular degeneration and other pathologies. The study hypothesis, never tested before, is that BT in cases with hemianopia will impact positively oculomotor control and visual acuity as it was proven to do in cases with macular degeneration.

Significance of the study

Vision is a major sensory input to the human brain. Half of the afferent neuronal fibers projecting to the brain originate from the eyes. Intact visual abilities are an important condition enabling us to orient ourselves in our world. Pambakian and Kennard 20 reported that 50% of all neurological admissions into hospitals in the United Kingdom are due to a stroke and 30% percent of them are reported to have hemianopia.

Numbers of hemianopic patients reported in the Czech Republic are similar and somewhat lower due to differences in diagnostics and classification of nosological units.21 Visual impairments are present in 20 to 40% of patients in neurological rehabilitation centers.

If brain visual plasticity is possible to be achieved from conventional vision training methods, specialized training with BT needs to be investigated as a tool to improve significantly a cortical visual disorder. There is need for simple and more effective visual training which could be used in LVR in large scale for hemianopia cases. Furthermore, BT needs to be evaluated in terms of quality of life (QoL) improvement to the patients.

The objectives set for this trial is to verify if BT impacts on oculomotor control in cases with hemianopia and results in better fixation stability, reading speed and QoL in those trained with BT.

ELIGIBILITY:
Inclusion Criteria:

* hemianopia cases previously diagnosed accordingly by microperimetry and other tests as needed
* 18-90 years old
* ability to follow the visual and auditory stimuli and training instructions

Exclusion Criteria:

* previous or current treatment for low vision rehabilitation
* ocular diseases
* other serious clinical conditions not related to the hemianopia physiopathology
* both eyes with media opacity that impairs microperimetry testing
* lack of ability to perform the tests and training

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 1 week post biofeedback
  ETDRS best corrected visual acuity
Fixation stability | 1 week post biofeedback
  As measure by the MAIA microperimeter at the BCEA 63% ellipse area.
Retinal sensitivity | 1 week post biofeedback
  Paracentral (2 central vertical columns) and total average in dB as measured by the MAIA microperimeter.
Reading speed | 1 week post biofeedback
  As measured with the MNRead charts
Near vision | 1 week post biofeedback
  Measured with the Colenbrander 100% charts
Quality of Life Questionnaire scores | 1 week post biofeedback
  As measured with the Massof - 48 questionnaire

SECONDARY OUTCOMES:
Stereopsis | 1 week post biofeedback
  As measured with the Frisby stereotest
Contrast Sensitivity | 1 week post biofeedback
  As measured with the F.A.C.T. test at 1m

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 2021 to 2026

REFERENCES:
- [Background] Kerkhoff G. Restorative and compensatory therapy approaches in cerebral blindness - a review. Restor Neurol Neurosci. 1999;15(2-3):255-71. PMID 12671237
- [Background] Bansal S, Han E, Ciuffreda KJ. Use of yoked prisms in patients with acquired brain injury: a retrospective analysis. Brain Inj. 2014;28(11):1441-6. doi: 10.3109/02699052.2014.919527. Epub 2014 Jun 9. PMID 24911923
- [Background] Nido MD, Markowitz SN. Vision rehabilitation with biofeedback training. Can J Ophthalmol. 2018 Jun;53(3):e83-e84. doi: 10.1016/j.jcjo.2017.11.003. Epub 2017 Dec 21. No abstract available. PMID 29784180
- [Background] Daibert-Nido M, Patino B, Markowitz M, Markowitz SN. Rehabilitation with biofeedback training in age-related macular degeneration for improving distance vision. Can J Ophthalmol. 2019 Jun;54(3):328-334. doi: 10.1016/j.jcjo.2018.10.016. Epub 2019 Apr 2. PMID 31109472
- [Background] Daibert-Nido M, Pyatova Y, Markowitz M, Markowitz SN. Visual outcomes of audio-luminous biofeedback training for a child with idiopathic nystagmus. Arq Bras Oftalmol. 2021 Mar-Apr;84(2):179-182. doi: 10.5935/0004-2749.20210026. PMID 33567015

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05397873/Prot_SAP_000.pdf